CLINICAL TRIAL: NCT04923386
Title: Effect of mRNA Based-Covid-19 Vaccine on Blood Glucose Levels Recorded by Continuous Glucose Monitoring in Patients With a History of Diabetes Mellitus Type I and Type II.
Brief Title: mRNA Based-Covid-19 Vaccine Effects on Blood Glucose Levels
Status: Completed | Type: Observational
Sponsor: Levenson, David I., M.D. (Individual)
Responsible Party: Principal Investigator, David I. Levenson, MD, Principal Investigator, Levenson, David I., M.D.
Other Study IDs: Macknofsky 1
Record Dates: First submitted 2021-06-06; First posted 2021-06-11 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1; Hyperglycemia; Vaccine Adverse Reaction
Keywords: mRNA Vaccine; Hyperglycemia; Hypoglycemia; Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1; COVID-19 Vaccine
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1; Hyperglycemia; Hypoglycemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diabetics who receive mRNA COVID-19 vaccine: Patients that have a history of Diabetes Mellitus Type I or Type II who received Pfizer-N-Biotech or Moderna mRNA COVID-19 vaccines
  Interventions: Other: None (not interventional)

INTERVENTIONS:
Other: None (not interventional) — This is not an intervention

SUMMARY:
To determine if patients with a history of Diabetes Mellitus Type I or II developed a change in blood glucose levels as reported on Continuous glucose monitoring devices (CGMS) within the first week following administration of each dose of the COVID-19 vaccine.

DETAILED DESCRIPTION:
A retrospective review of all patient data from the Dexcom and Libre CGMS devices available at a single site, solo endocrinology practice will be obtained. This data will include fasting morning glucose, postprandial glucose, and daily glucose area under the curve for seven days following vaccination administration, as well as daily glucose area under the curve seven days prior to vaccine administration that will be used as a control. Patients >=18 y/o with a history of Diabetes Mellitus Type I or Type II will be selected. Brand of vaccine administered (Moderna or Pfizer-BioNTech) and the change in average blood glucose, peak blood glucose, and percentage of time spent in normal range as well as above average range of blood glucose level following vaccine administration will be assessed. Patients will fill out a visual analog symptom scale based on how symptomatic and uncomfortable they were following each dose of the COVID-19 vaccine. Patients will describe side effects that they experienced following each dose of the COVID-19 vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Diabetes Mellitus Type I or Type II
* Received the Moderna COVID-19 vaccine or Pfizer-BioNTech COVID-19 vaccine

Exclusion Criteria:

* Patients <18y/o.
* Patients that did not receive a COVID-19 vaccine.
* Patients who did not have a CGMS downloaded for a week prior and a week after vaccination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All eligible patients in the PI's database.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Change in AUC glucose level above expected baseline | 7 days
  Change in area under the curve glucose level above expected baseline

SECONDARY OUTCOMES:
Change in peak glucose level above expected baseline | 7 days
  Change in peak glucose level above expected baseline
Change in fasting blood glucose levels above expected baseline | 7 days
  Change in fasting blood glucose levels above expected baseline

CONTACTS AND LOCATIONS:
Overall Officials: David I Levenson, M.D., Principal Investigator — East Coast Medical Associates
Locations (1):
- East Coast Medical Associates, Boca Raton, Florida, United States

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared.